CLINICAL TRIAL: NCT02405052
Title: A Prospective Cohort Study to Refine and Validate the Panic Screening Score for Identifying Panic Attacks Associated With Unexplained Chest Pain in the Emergency Department
Brief Title: Validation of the Panic Screening Score in Patient With Unexplained Chest Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CISSS de Chaudière-Appalaches (Other Government)
Responsible Party: Principal Investigator, Guillaume Foldes-Busque, Chercheur, CISSS de Chaudière-Appalaches
Other Study IDs: 286934
Record Dates: First submitted 2015-03-29; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Noncardiac Chest Pain; Panic Attack
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Patients: Emergency department patients with unexplained chest pain
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Validation of the Panic Screening Score

SUMMARY:
Panic-like anxiety ( panic attacks with or without panic disorder), a highly treatable condition, is the most prevalent condition associated with unexplained chest pain in the emergency department. Panic-like anxiety may be responsible for a significant portion of the negative consequences of unexplained chest pain, such as functional limitations and chronicity. However, more than 92% of panic-like anxiety cases remain undiagnosed at the time of discharge from the emergency department. The 4-item Panic Screening Score questionnaire was derived in order to increase the identification of panic-like anxiety in emergency department patients with unexplained chest pain.

The goals of this prospective cohort study are to (1) refine the Panic Screening Score; (2) validate the revised version of the Panic Screening Score; (3) measure the reliability of the revised version of the Panic Screening Score and (4) assess the acceptability of the instrument among emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

Presenting unexplained chest pain as defined by:

* the absence of an identifiable cause (e.g., pneumothorax,pneumonia),
* the absence of chest trauma,
* the absence of new malignant cardiac arrhythmia, and
* a score of 2 or less on the modified version of the thrombolysis in myocardial infarction score.

Exclusion Criteria:

* presence of a terminal illness;
* presence of a severe communication problem that could interfere with the administration of the questionnaire;
* presence of a psychotic state, a major cognitive deficit or other condition that could invalidate the interview;
* being legally incompetent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the emergency department
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the Panic Screening Score | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Foldes-Busque, Ph.D, Principal Investigator — Centre hospitalier affilié universitaire de Lévis
Locations (1):
- Centre de recherche, CSSS Alphonse-Desjardins, Centre hospitalier affilié universitaire de Lévis, Lévis, Quebec, Canada

REFERENCES:
- [Background] Foldes-Busque G, Denis I, Poitras J, Fleet RP, Archambault P, Dionne CE. A prospective cohort study to refine and validate the Panic Screening Score for identifying panic attacks associated with unexplained chest pain in the emergency department. BMJ Open. 2013 Oct 25;3(10):e003877. doi: 10.1136/bmjopen-2013-003877. PMID 24163208